CLINICAL TRIAL: NCT01475565
Title: Insulin Resistance Before and During Pregnancy in Women With PCOS
Brief Title: Insulin Resistance Before and During Pregnancy in Women With Polycystic Ovary Syndrome
Status: Terminated | Type: Observational
Why Stopped: Only 2 participants were enrolled
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: HM13733
Record Dates: First submitted 2011-11-08; First posted 2011-11-21 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Polycystic Ovary Syndrome; Insulin Resistance; Insulin Sensitivity; Obesity; Pregnancy
Keywords: polycystic ovary syndrome (PCOS); insulin sensitivity; insulin resistance; gestational diabetes; pregnancy; estrogen; glucose intolerance; obesity; ovulatory disorder; racial differences; hyperandrogenism
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance; Obesity; Diabetes, Gestational; Glucose Intolerance; Hyperandrogenism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * blood sample
  * blood sample sample for DNA
  * fasting plasma for insulin, glucose, sex steroids (testosterone, androstenedione, DHEA-sulfate, estradiol, estrone, progesterone), sex hormone-binding globulin and estrogen metabolites
  * blood sample for oral glucose tolerance test
  * urine for estrogen metabolites
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- African-American women: Observational study--no intervention
- Caucasian women: Observational study--no intervention

SUMMARY:
The polycystic ovary syndrome (PCOS) affects about 10% of reproductive-age women. Women with PCOS are at a higher risk of gestational diabetes, which may lead to more pregnancy complications. It is unknown if there are factors that may predict which women are more at risk.

The goal of this study is to evaluate the risk factors of gestational diabetes, such as dietary and physical activity factors, race, and how the body handles its own hormones during pregnancy. Our long term goal is to contribute in finding ways to successfully prevent gestational diabetes.

DETAILED DESCRIPTION:
The polycystic ovary syndrome is the leading cause of female infertility in the United States. The disorder affects approximately 6-10% of women of reproductive age. Insulin is a hormone that helps the body to take up sugar from the bloodstream. It is widely accepted that "insulin resistance" may be responsible for the polycystic ovary syndrome. Women are insulin resistant when their bodies do not respond to insulin's action to handle sugar as they normally should. Because of this insulin resistance, when women with the polycystic ovary syndrome become pregnant, they are at a higher risk of developing gestational diabetes. Gestational diabetes carries risk to both the mother and the baby. The purpose of this study is to determine whether certain factors in women with the polycystic ovary syndrome are linked to risk of gestational diabetes. We propose to look at demographic factors, as well as the body's handling of estrogen (a female hormone present in high quantities during pregnancy) in this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PCOS prior to pregnancy
* 18-40 years of age
* Documented BMI 30-40 kg/m2 (within 3 months prior to pregnancy or within 8 weeks of gestation)
* Either of Caucasian or African-American decent by self report.
* Pregnant or attempting pregnancy

Exclusion Criteria:

* Preexisting Diabetes (impaired glucose tolerance will not be an exclusion criterion because of the high prevalence of impaired glucose tolerance in the PCOS population).
* Hemoglobin < 8 or hemoglobin <10 with symptoms of anemia.
* Use of tobacco, alcohol or illicit substances.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants will be recruited from clinics in/near Richmond, VA.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2013-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change from Gestation Week 12-14 in Estrogen Metabolites at Gestation Week 32-34 | Gestation weeks 12-14, 24-26, and 32-34
Change from Gestation Week 12-14 in Insulin Sensitivity at Gestation Week 32-34 | Gestation weeks 12-14, 24-26, and 32-34

SECONDARY OUTCOMES:
Change from Gestation Week 12-14 in Fasting Insulin at Gestation Week 32-34 | Gestation weeks 12-14, 24-26, and 32-34
Change from Gestation Week 12-14 in Fasting Glucose at Gestation Week 32-34 | Gestation weeks 12-14, 24-26, and 32-34
Change from Gestation Week 12-14 in Areas-under-the-response-curve of Insulin at Gestation Week 32-34 | Gestation weeks 12-14, 24-26, and 32-34
Change from Gestation Week 12-14 in Areas-under-the-response-curve of Glucose at Gestation Week 32-34 | Gestation weeks 12-14, 24-26, and 32-34
Change from Gestation 12-14 in Matsuda Insulin Sensitivity Index at Gestation Week 32-34 | Gestation weeks 12-14, 24-26, and 32-34
Change from Gestation Week 12-14 in Insulin Secretory Response at Gestation Week 32-34 | Gestation weeks 12-14, 24-26, and 32-34
Change from Gestation Week 12-14 in Macronutrients at Gestation Week 32-34 | Gestation weeks 12-14, 24-26, and 32-34
Change from Gestation Week 12-14 in Urinary Estrogen Metabolites at Gestation Week 32-34 | Gestation weeks 12-14, 24-26, and 32-34
Change from Gestation Week 12-14 in Body Weight at Gestation Week 32-34 | Gestation weeks 12-14, 24-26, and 32-34
Change from Gestation Week 12-14 in Physical Activity at Gestation Week 32-34 | Gestational week 12-14, 24-26, 32-34

CONTACTS AND LOCATIONS:
Overall Officials: Kai Cheang, Pharm. D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University Medical Center, Richmond, Virginia, United States